CLINICAL TRIAL: NCT04549623
Title: The Effect of A Novel End-Tidal Carbon Dioxide Monitoring Device for Sedation During Endoscopic Ultrasonography-Guided Fine Needle Aspiration
Brief Title: End-Tidal Carbon Dioxide Monitoring Device for Sedation During Endoscopic Ultrasonography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Jia-feng Wang, Principal Investigator, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ETCO2-MDS
Record Dates: First submitted 2020-08-31; First posted 2020-09-16 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Endoscopic Ultrasonography; Sedation; Monitoring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ETCO2 (Experimental): Novel end-tidal carbon dioxide monitoring device is used for sedation.
  Interventions: Device: Novel end-tidal CO2 monitoring device
- Group Reg (Experimental): Peripheral oxygen saturation (SpO2) and respiratory motion are regularly monitored during sedation.
  Interventions: Device: SpO2 and respiratory motion monitoring

INTERVENTIONS:
Device: Novel end-tidal CO2 monitoring device — Apart from SpO2 and respiratory motion monitoring, the EtCO2 monitoring device is used to detect CO2 from nose and mouth simultaneously.
  Arms: Group ETCO2
Device: SpO2 and respiratory motion monitoring — Finger SpO2 and ECG-based respiratory motion monitoring are used during operation.
  Arms: Group Reg

SUMMARY:
To meet the needs of both operators and patients, moderate and deep sedation has been widely used in digestive endoscopy, which is invasive and painful. With its pleasant effects, sedation has complications nevertheless. And respiratory depression is the most common one, which makes respiratory monitoring significant. SpO2 and respiratory motion are regularly monitored without satisfying timeliness or sensitivity. Capnography with current device is only able to detect either oral or nasal breathing. The present study was designed to test the effect of the investigator's modified End-Tidal Carbon Dioxide (ETCO2) monitoring device for sedation during endoscopic ultrasonography-guided fine needle aspiration.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for ultrasonography-guided fine needle aspiration
* Adult patients aged 18 to 65 years
* American Society of Anesthesiologists (ASA) Physical Status Classification I-III
* Subjects provide informed consent

Exclusion Criteria:

* Full stomach or upper gastrointestinal tract obstruction
* Baseline pulse oximetric saturation (SpO2) <95% while breathing room air
* Obesity （BMI≥28kg/m2）or anticipated difficult airway
* Cardiovascular or cerebrovascular events within 3 months
* Pregnancy
* Chronic opioid user
* Allergic to anesthetics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2020-09-27 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Peripheral oxygen saturation | Across the sedation, assessed up to 2 hours
  Peripheral oxygen saturation is measured by pulse oximetry and hypoxemia is defined as SpO2≤91%

SECONDARY OUTCOMES:
Arterial pO2 and pCO2 | 30 minutes after initiation of the sedation
  The results of arterial blood gas measurements including partial pressure of oxygen (pO₂) and carbon dioxide (pCO₂)
The numbers of the times of body movement | From the completion of sedation to the completion of endosonography procedure, assessed up to 2 hours
  The numbers of the times of any body movement across the procedure
Incidence of hypertension and hypotension | From the completion of sedation to the completion of endosonography procedure, assessed up to 2 hours
  Hypertension or hypotension is defined as an increase or decrease in systolic blood pressure ≥20% compared to baseline values
Recovery time | After termination of the sedation medication, assessed up to 2 hours
  Duration of the recovery from sedation
Total dosage of propofol | Across the sedation, assessed up to 2 hours
  The patients are induced with 1.5~2.5mg/kg and maintained with 6~10mg/(kg•h) propofol. A propofol bolus dose range 0.2~0.5 mg/kg will be administered when needed.
Satisfaction score of the patients and endosonographers | Across the procedure, assessed up to 2 hours
  Satisfaction score of the patients and endosonographers regarding to the sedation quality measured by a 0-100 visual analogue scale (VAS). 100 refers to the highest satisfaction degree while 0 refers to the worst satisfaction degree.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Anesthesiology, Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided